CLINICAL TRIAL: NCT05393050
Title: Efficacy and Safety of Colquhounia Root Tablet in Patients With Rheumatoid Arthritis：A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Colquhounia Root Tablet in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Quan Jiang (Other)
Responsible Party: Sponsor-Investigator, Quan Jiang, chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-001P6A01
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Colquhounia Root Tablet; Methotrexate; Randomized controlled trial
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colquhounia Root Tablet plus methotrexate (MTX) (Active Comparator): Colquhounia Root Tablet 0.9g tid and methotrexate (MTX) 10 mg oncea week for the first 12 weeks，Colquhounia Root Tablet 0.54g tid and methotrexate (MTX) 10 mg once a week for the after 12 weeks.
  Interventions: Drug: Colquhounia Root Tablet; Drug: Methotrexate tablets
- placedo of Colquhounia Root Tablet plus methotrexate (MTX) (Placebo Comparator): placedo of Colquhounia Root Tablet 0.9g tid and methotrexate (MTX) 10 mg oncea week for the first 12 weeks，placedo of Colquhounia Root Tablet 0.54g tid and methotrexate (MTX) 10 mg once a week for the after 12 weeks.
  Interventions: Drug: Methotrexate tablets

INTERVENTIONS:
Drug: Colquhounia Root Tablet — Colquhounia Root Tablet is a tripterygium preparation
  Arms: Colquhounia Root Tablet plus methotrexate (MTX)
Drug: Methotrexate tablets — Methotrexate is a drug used to treat rheumatoid arthritis

SUMMARY:
This study is a multi-center, randomized, double-blinded, controlled trial with two parallel arms. The aim of the study is to evaluate whether Colquhounia Root Tablet combined with methotrexate (MTX) might be better than MTX alone for patients with active rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

1. Subject understood the whole process of the trial and signed the informed consent voluntarily.
2. Subject has had a confirmed diagnosis of rheumatoid arthritis according to 2010 ACR/EULAR RA classification criteria.
3. Subjects aged between 45-70years who were the males without fertility requirements or menopausal women.
4. Subject has a DAS28 CRP disease activity score greater than 2.6 and less than 5.1.
5. Subject did not participate in any drug trials within 1 month before enrollment.

Exclusion Criteria:

1. Pregnant women, women planning to become pregnant or breastfeeding.
2. Severe systemic involvement, such as severe pericardial effusion, interstitial lung disease, renal tubular acidosis, autoimmune liver disease.
3. Active liver disease or abnormal liver function, ALT and AST are more than 1.5 times the upper limit of normal.
4. Renal impairment, serum creatinine greater than the upper limit of normal.
5. Bone marrow hematopoietic dysfunction, peripheral blood leukocytes <3.0×109/L, or definite anemia (hemoglobin less than 80g/L), or platelets <80×109/L, or other blood system diseases.
6. Active gastric and duodenal ulcers.
7. Uncontrolled severe hypertension, metabolic diseases.
8. malignant tumors.
9. Acute and/or chronic infectious diseases.
10. Severe cardiac arrhythmia found on electrocardiogram.
11. Mental illness, history of alcoholism, drug or other substance abuse.
12. Diagnosed with other connective tissue disease.
13. Those who have used immunosuppressants, biological agents, Colquhounia Root Tablet or drugs containing Tripterygium wilfordii within 1 month before enrollment.
14. Those who have previously used methotrexate or preparations containing tripterygium wilfordii for 12 weeks or more ,but their condition is not under control.
15. Adverse reactions have occurred in the past using Colquhounia Root Tablet or drugs containing Tripterygium wilfordii.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of ACR20 | week 24
  Percentage of Participants With American College of Rheumatology 20% (ACR20)

SECONDARY OUTCOMES:
Percentage of ACR50 | week 24
  Percentage of Participants With American College of Rheumatology 50% (ACR50)
Percentage of ACR70 | week 24
  Percentage of Participants With American College of Rheumatology 70% (ACR70)
DAS28-ESR | week 24
  28-joint disease activity score
Chinese Patient-reported Activity Index with RA scale (PRO) | week 24
  Patient-Reported Outcomes Scale,The self-rating scale consists of 12 items,Each item was rated 0, 1, 2 and 3 on the scale of asymptomatic to aggravating symptoms, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No